CLINICAL TRIAL: NCT00410436
Title: Resistance Exercise in Already-active Diabetic Individuals (READI) Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005301-01H; 2005783 (Other: OHREB)
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes
Keywords: Type 1 Diabetes; Resistance Exercise; Aerobic Exercise
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resistance Training Group (Experimental): Resistance Training (R) 3X/week progressing to 3 sets, 8 repetitions of 8 exercises at the maximum load that can be lifted 8 times in a controlled manner, maintaining proper form (8RM).
  Interventions: Behavioral: Resistance Exercise
- Control Group (Active Comparator): Subjects will not be performing resistance exercise but will continue performing aerobic exercise at the same volume, duration and intensity as they did at baseline.
  Interventions: Behavioral: Resistance Exercise

INTERVENTIONS:
Behavioral: Resistance Exercise — Subjects demonstrating adequate compliance during the run-in period will then be randomized in equal numbers to Resistance Training (R) 3X/week progressing to 3 sets, 8 repetitions of 8 exercises at the maximum load that can be lifted 8 times in a controlled manner, maintaining proper form (8RM), or waiting-list control (C).
  Other Names: non applicable

SUMMARY:
The purpose of the READI tiral is to examine the effects of resistance training (weight training) on the blood sugar control of aerobically active individuals with Type 1 Diabetes.

DETAILED DESCRIPTION:
Background: Juvenile-onset type 1 (insulin-dependent) diabetes is associated with a 15 year reduction in life expectancy, primarily due to cardiovascular disease (CVD). Poor blood glucose (glycemic) control, reflected in elevated hemoglobin A1c (HbA1c) is a major risk factor for diabetes complications; each 1% absolute reduction in HbA1c leads to a 15-20% reduction in risk of a major cardiovascular event, and a 25-37% reduction in risk of microvascular disease. Exercise is appealing as a potential non-pharmacological intervention to improve glycemic control. However, while aerobic exercise (e.g. walking, running) improves insulin sensitivity, most published studies found that aerobic exercise did not improve glycemic control in type 1 diabetes. This paradoxical finding is likely due to the tendency of type 1 diabetic individuals to decrease their insulin doses and/or increase carbohydrate intake more than necessary in order to avoid exercise-induced hypoglycemia. In comparison to aerobic exercise, the smaller acute rise in glucose uptake associated with resistance exercise may offer the metabolic benefits of exercise while minimizing risk of exercise-induced hypoglycemia. Only two small published studies (n=8 and 10; men only) evaluated resistance exercise (weight lifting or exercises with weight machines) in type 1 diabetes, but their results were promising. In a crossover trial, glycemic control was significantly better during resistance training than during non-exercise control (HbA1c 5.8% versus 6.9%; absolute difference 1.1%). In a before-after study, combined aerobic and resistance exercise reduced absolute HbA1c by 0.96%. People with type 1 diabetes who already do regular aerobic exercise would likely be open to starting an additional form of exercise if it were proven to improve glycemic control. We therefore wish to evaluate the incremental effect of resistance training on HbA1c in already-aerobically-active type 1 diabetic individuals in a randomized, controlled trial.

Primary research question: In type 1 diabetic individuals who already engage in regular aerobic exercise, does adding a 6-month resistance training program result in improved glycemic control as reflected in reduced HbA1c compared to aerobic training alone?

Secondary research questions: In type 1 diabetic individuals who already do regular aerobic exercise, does adding a 6-month resistance training program have favourable effects on body composition, non-traditional and traditional CVD risk factors, and quality of life vs. aerobic exercise alone?

Exploratory research questions: What is the incremental effect of resistance training on insulin requirements and frequency of hypoglycemia? Do changes in glycemic control, body composition, or quality of life during the resistance training intervention predict exercise participation during the subsequent 6 months? How cost-effective is it to add the resistance training program?

Methods: Type 1 diabetic subjects aged ≥16 yr who perform aerobic exercise ≥3 times per week but not resistance exercise, will be recruited at three centres (Ottawa, Toronto and Calgary). They will first enter a 5-week run-in period, including 3X/week supervised low-intensity resistance exercise training in weeks 2-5. During run-in, in addition to verifying adherence to the exercise program, intense efforts will be made to optimize diabetes care including frequent interaction with the study diabetes nurse/educator and dietitian, intensification and adjustment of insulin therapy. Subjects attending ≥80% of the exercise sessions and demonstrating good compliance with diabetes care during run-in will then be randomized to either resistance training or waiting list control for weeks 6-26; in either case they will continue aerobic exercise at their usual volume and intensity with support from an Exercise Specialist, use pedometers and report exercise in activity logs. Resistance exercise training in the intervention group will progress to 3 sets of 8 reps of 8 exercises at 8RM (maximum weight that can be lifted 8 times while maintaining proper form). Background diabetes care will be provided throughout, in a protocolized manner for both exercise and control subjects, with all insulin adjustments done by study research staff.

Significance: Reduced risk of long-term complications of type 1diabetes is tightly linked to better glycemic control, which is often difficult to achieve. This study will provide valuable information regarding the extent to which resistance exercise can improve glycemic control and other important risk factors for complications in people with type 1 diabetes who are already aerobically active.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus as defined by the 2003 CDA guidelines with duration ≥1 year, requiring insulin therapy starting within one year of diagnosis and continuously thereafter.
* Male or female, age ≥16 years, HbA1c 0.066-0.099 (normal non-diabetic range 0.040-0.060).
* Habitual performance during the previous 4 months of exercise ≥3 times per week, including at least 90 minutes per week of vigourous aerobic exercise (of sufficient intensity to cause sweating; e.g. jogging, soccer, basketball, racquet sports), and/or ≥150 minutes per week of aerobic exercise of at least moderate intensity (e.g. brisk walking, moderate-paced bicycling) but no resistance training. Subjects must agree to maintain their habitual volume and intensity of aerobic activity during run-in and intervention periods, minimizing variation due to seasons, but they will be permitted to vary specific exercises chosen.
* Willingness and ability to work closely with the study physicians, nurse and dietitian and follow their recommendations for insulin therapy and adjustments of diet.

Exclusion Criteria:

* Participation during the previous 4 months in any resistance training.
* Hypoglycemia unawareness, or severe hypoglycemia requiring assistance from another person within the previous 3 months
* "Brittle" diabetes, characterized by frequent and unpredictable hypoglycemia (even if not requiring assistance from others) and hyperglycemia.
* Restrictions in physical activity due to disease: intermittent claudication, severe peripheral neuropathy or active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis.
* Known or suspected clinically significant gastroparesis.
* Body mass index >35 kg/m2, or weight >147 kg (exceeding capacity of DEXA or CT scanners)
* Fasting serum c-peptide 0.2 nmol/l.
* Increase or decrease of 5% of body weight during the previous two months.
* An expected requirement within the subsequent 6 months for medications (other than insulin) that will affect glucose metabolism (e.g. corticosteroids).
* If age<18 yr, linear growth of 1cm during the previous year.
* Significant renal disease: serum creatinine 200 mEq/l. or proteinuria >1 g/24 hours.
* Uncontrolled hypertension: BP >150 mm Hg systolic or >95 mm Hg diastolic in a sitting position.
* Other illness, judged by the patient or investigators to make participation in this study inadvisable.
* Cognitive deficit resulting in inability to understand or comply with instructions.
* Pregnancy at the start of the study, or intention to become pregnant in the next year.
* Inability to communicate in English or French.
* Ischemic ECG changes during baseline maximal cardiopulmonary stress test, unless subsequently cleared for participation by a cardiologist after appropriate investigation.
* Low aerobic fitness: Aerobic fitness more than 15% below the mean for age and gender, based on baseline maximal treadmill exercise test. This criterion is included in order to reduce likelihood of candidates entering the trial by exaggerating their habitual activity. Very few people engaging in regular aerobic activity would have such low treadmill performance.
* Unwillingness to sign informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-10; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6-months
  Change in HbA1c from pre and post-intervention

SECONDARY OUTCOMES:
body composition,LDL particle diameter,apolipoprotein B (Apo-B) | 6-months
  measured pre and post exercise intervention
apolipoprotein A1 (Apo-A1,Apo-B/Apo-A1 ratio,urinary albumin excretion | 6-months
  measured pre and post exercise intervention
serum C-reactive protein, | 6-months
  measured pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ron Sigal, MD, Study Chair — OHRI
Locations (3):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - Ottawa Health Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario